CLINICAL TRIAL: NCT05573932
Title: The Effects of a Gamified Rehabilitation Protocol Compared to an At-Home Exercise Packet in Individuals With Low Back Pain
Brief Title: Gamified Rehab vs Take-home Packet Rehab for Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00004656
Record Dates: First submitted 2022-09-26; First posted 2022-10-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Non-specific Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized into the two separate groups using a random number generator and allocation will be concealed in opaque envelopes prior to data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leaderboard group (Experimental): The group that has access to weekly leaderboards and on-demand videos.
  Interventions: Other: Leaderboard
- Take-home packet group (Active Comparator): The group that has access to paper take-home packets.
  Interventions: Other: Take-home packet

INTERVENTIONS:
Other: Leaderboard — De-identified leaderboard showing average durations of exercises completed by all participants in leaderboard group.
  Arms: Leaderboard group
Other: Take-home packet — Take-home packet of exercises.
  Arms: Take-home packet group

SUMMARY:
Two groups with non-specific low back pain will be completing the same exercise protocol. The leaderboard group will have a gamified experience and the take-home packet group will be using a paper take-home packet. Outcomes will be measured at 3 weeks, 6 weeks, with pain and disability also being measured at 12 and 18 months.

DETAILED DESCRIPTION:
There will be two groups in this study, the leaderboard group, and the take-home packet group. The leaderboard group and the take-home packet group will be completing the same exercise program throughout the 6-weeks. The exercises included the plank, side plank (left and right side), foot elevated (left and right side), dead bug and bird dog exercise until discontinuation. The exercises will increase with repetitions every two weeks and that outline is listed below in procedures involved. The leaderboard group will have on demand video access to the exercises and the take-home packet group will have a take-home packet. The leaderboard group will also be receiving weekly leaderboards of average and top exercise durations of the leaderboard group participants. The audio description of exercise in the on-demand video group is the same script as the written description in the take-home packet.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18-45 years old
* Biological sex of Male or Female
* Self-reported low back pain within the previous 6 months or greater than 3 episodes within the past 3 years

Exclusion Criteria:

* Must not be currently seeing and or receiving care from an athletic trainer, physical therapist, or other rehabilitation specialist in the previous 6 months
* Must not have low back pain conditions such as lumbar spondylosis, herniated disc, spondylolisthesis, previous spine surgery, currently pregnant, experiencing neurological symptoms or other muscular abnormalities
* Unable to assume the exercise starting position
* Current use of lidocaine patches or prescription pain medicine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain | Change from baseline to 3 weeks
  Assessed by the numeric pain rating scale
Change in pain | Change from baseline to 6 weeks
  Assessed by the numeric pain rating scale
Change in pain | Change from baseline to 12 months
  Assessed by the numeric pain rating scale
Change in pain | Change from baseline to 18 months
  Assessed by the numeric pain rating scale
Change in Disability | Change from baseline to 3 weeks
  Assessed with the Oswestry Disability Index
Change in Disability | Change from baseline to 6 weeks
  Assessed with the Oswestry Disability Index
Change in Disability | Change from baseline to 12 months
  Assessed with the Oswestry Disability Index
Change in Disability | Change from baseline to 18 months
  Assessed with the Oswestry Disability Index
Adherence | Change from baseline to 3 weeks
  Assessed by the exercise adherence rating scale
Adherence | Change from baseline to 6 weeks
  Assessed by the exercise adherence rating scale
Change in Muscle thickness of the lateral abdominal wall | Change from baseline to 6 weeks
  Assessed with ultrasound during static positions and exercise starting positions

CONTACTS AND LOCATIONS:
Locations (1):
- READY Laboratory, Education Complex, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devorski L, Suppiah A, Fukuda DH, Stout J, Ingersoll CD, Mangum LC. Gamified delivery of at-home rehabilitation for individuals with nonspecific low back pain: a randomized controlled trial. Disabil Rehabil. 2025 Mar;47(6):1416-1422. doi: 10.1080/09638288.2024.2368694. Epub 2024 Jun 20. PMID 38899776

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT05573932/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT05573932/ICF_001.pdf